CLINICAL TRIAL: NCT04072731
Title: SREBP1 as a Potential Biomarker Promotes Cell Proliferation and Invasion in Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: People's Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Zhi Li, Xiangya Hospital, Central South University, People's Hospital of Zhengzhou University
Other Study IDs: SBQLL-2016-015
Record Dates: First submitted 2018-01-16; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer; SREBP1
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Iodine-131

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Tissue samples were snap-frozen and stored in liquid nitrogen immediately after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- thyroid cancer: the thyroid cancer was determined by the the Pathology Department based on the pathological evidence.
  Interventions: Other: pathologic
- the adjacent thyroid tissues: the adjacent thyroid tissues was collected from the tissue that 3 centimeters from the thyroid cancer.
  Interventions: Other: pathologic

INTERVENTIONS:
Other: pathologic — All the enrolled patients were treated with whole resection and diagnosed by the Pathology Department based on the pathological evidence.
  Other Names: radioiodine

SUMMARY:
In this study, the investigators detected the expression of SREBP1 in thyroid cancer tissues, explored the biological functions of SREBP1 in thyroid cancer cells.

DETAILED DESCRIPTION:
qRT-PCR and immunohistochemistry were used to detect the expression of SREBP1 in 96 pairs thyroid cancer tissues and the adjacent normal tissues. The following methods, including the MTS, colony-forming assay, flow cytometry and hoechst staining were used to detect the biological function of thyroid cancer cells based on SREBP1 interference or not.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of thyroid cancer Reciving thyroidectomy surgery No experience of radiation therapy Nice treatment compliance and follow-up regularly

Exclusion Criteria:

Prior history of malignancy ; Radiotherapy history, chemotherapy history; Serious concomitant diseases ; Chronic renal insufficiency and liver dysfunction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: all of this patients were recruited from the Affiliated Cancer Hospital of Xiangya Medical School
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-01-16 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
progression-free survival | average 5 years
  disease recurrent of progression

SECONDARY OUTCOMES:
theraputic efficacy | average 18 months
  According to the ATA guideline, patients were divided into four group, including excellent response (ER),indeterminate response (IDR), biochemical incomplete response (BIR), structural incomplete response (SIR) after surgery and radioiodine treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Li, Prof., Principal Investigator — Central South University
Locations (1):
- the Affiliated Cancer Hospital of Xiangya Medical School, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No